CLINICAL TRIAL: NCT04980196
Title: Is Urodynamic Study an Essential Step in Preoperative Evaluation of Women With Pelvic Organ Prolapse With Urinary Tract Dysfunction: Prospective Comparative Study
Brief Title: Is Preoperative Urodynamics Essential for Women With Pelvic Organ Prolapse
Acronym: urodynaemics
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mervit Sersy, Assistant professor, Alexandria University
Other Study IDs: 0304824
Record Dates: First submitted 2021-07-18; First posted 2021-07-28 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Urogenital Prolapse
Keywords: pelvic organ prolapse,; Urodynamics
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- (1) URODYNAEMICS GROUP: 30 patients allocated for group (1) had been thoroughly evaluated by history and examination. A standardized questionnaire was obtained to evaluate the symptoms of stress urinary incontinence, urge urinary incontinence and obstructive symptoms. Clinical staging of pelvic organ prolapse by POP Q Staging .Ultrasound examination had been also carried out to rule out any pelvic pathology. Patients had completed a 3-day bladder diary (frequency volume chart) to assist in arriving at an urodynamic diagnosis. Urinalysis was performed. And to urodynamic studies were performed before surgical intervention and then corrective procedures for POP had been done uroflowmetry and cystometry. All participants were followed-up with same questionnaire and clinical examination after 12 weeks post -operatively
  Interventions: Diagnostic Test: urodynaemic studies
- (2)NON URODYNAMICS GROUP: 30 patients allocated for group (2) had been thoroughly evaluated by history and examination. A standardized questionnaire was obtained to evaluate the symptoms of stress urinary incontinence, urge urinary incontinence and obstructive symptoms. Clinical staging of pelvic organ prolapse by POP Q Staging .Ultrasound examination had been also carried out to rule out any pelvic pathology. Patients had completed a 3-day bladder diary (frequency volume chart) to assist in arriving at an urodynamic diagnosis. Urinalysis was performed and then corrective procedures for POP had been done.All participants were followed-up with same questionnaire and clinical examination after 12 weeks post-- operatively

INTERVENTIONS:
Diagnostic Test: urodynaemic studies — The Urodynamic studies carried out were : uroflowmetry and cystometry. The Uroflowmetry was performed by the gravimetric method Detrusor over activity was diagnosed when the patient has involuntary detrusor contractions during filling with or without leakage which may be spontaneous or provoked,
  Groups: (1) URODYNAEMICS GROUP

SUMMARY:
urodynamic investigation when added in the diagnostic work-up of women with lower urinary tract dysfunction with POP is debatable.

This study was planned to determine the usefulness of preoperative urodynamic study in improving urological outcome following surgery in women with pelvic organ prolapse and urinary tract dysfunction.

DETAILED DESCRIPTION:
60 patients, fulfilled the selection criteria were counseled and informed about the trial protocol and a written consent according to declaration of Helsinki was signed. Participants were randomly assigned following simple randomization procedures (computerized random numbers) to group (1) or group (2). Each group consisted of 30 patients. All participants had been thoroughly evaluated by history and examination. A standardized questionnaire was obtained to evaluate the symptoms of stress urinary incontinence, urge urinary incontinence and obstructive symptoms. Clinical staging of pelvic organ prolapse by POP Q Staging. Ultrasound examination had been also carried out to rule out any pelvic pathology. Patients had completed a 3-day bladder diary (frequency volume chart) to assist in arriving at an urodynamic diagnosis. Urinalysis was performed. Only patients allocated for group 1 were subjected to urodynamic studies before surgical intervention and then corrective procedures for POP had been done .The Urodynamic studies carried out were : uroflowmetry and cystometry. The Uroflowmetry was performed by the gravimeter method, where maximum flow rate, average flow rate, voided volume and residual urine was measured. Maximum flow rate ≤15 ml/sec, and/or residual urine of more than 50 ml or 10% of voided volume in a bladder filled with a minimum of 150 ml was taken as cut off to detect abnormal voiding. Cystometric parameters which indicated normal bladder function were first desire to void between 150 and 200 ml, capacity (taken as strong desire to void) of greater than 400 ml, detrusor pressure rise on filling of less than 15 mm H2O per 500 ml infused, absence of detrusor contractions, no leakage on coughing, no significant pain on filling and finally a detrusor pressure rises on voiding (maximum voiding pressure) of less than 50 cm H2O, with a peak flow rate of more than 15 ml/s for a voided volume over 150 ml. Urodynamic stress incontinence was diagnosed when urethral leakage was seen with increased abdominal pressure, in the absence of detrusor contractions. Detrusor over activity was diagnosed when the patient has involuntary detrusor contractions during filling with or without leakage which may be spontaneous or provoked. All participants were followed-up with same questionnaire and clinical examination after 12 weeks post operatively.

ELIGIBILITY:
Inclusion Criteria:

- pelvic organ prolapse associated with lower urinary tract dysfunction.

Exclusion Criteria:

* are those who had previous surgery for urinary incontinence, or experienced neurological disorder such as multiple sclerosis or spinal cord injuries were not included. Or had complicated medical disease that made the patient unfit for anesthesia.

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: performed in Shatby Maternity University hospital, which is considered the largest hospital in Alexandria city in Egypt offering obstetrical and gynecological services for more than three millions females
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
urological outcome following surgery in women with pelvic organ prolapse and urinary tract dysfunction. | 3months
  persistence of urinary incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Mervat AM Elsersy, MD, Principal Investigator — Alexandria University
Locations (1):
- Shatby Maternity University Hospital, Alexandria, El-Khartoum Square, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication
Access Criteria: Researcher of the same institution
URL: http://www.med.alexu.edu.eg